CLINICAL TRIAL: NCT03252340
Title: Observational Study to Evaluate the Safety of ADSTEM Injection in Patients With Moderate to Severe Subacute and Chronic Atopic Dermatitis
Brief Title: Safety of ADSTEM Injection in Patients With Moderate to Severe Subacute and Chronic Atopic Dermatitis
Status: Completed | Type: Observational
Sponsor: EHL Bio Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: AD-CP-17-1; 30902 (Other Grant/Funding Number: Republic or Korea Ministry of Food and Drug Safety)
Record Dates: First submitted 2017-08-08; First posted 2017-08-17 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Drug: ADSTEM Inj.: Participants in Phase I clinical trials treated with ADSTEM Inj.
  Interventions: Drug: ADSTEM Inj.

INTERVENTIONS:
Drug: ADSTEM Inj. — 1. ADSTEM Inj. 1.0x10^8 mesenchymal stem cells as an intravenous infusion once in Phase I clinical trial.
  2. ADSTEM Inj. 3.0x10^8 mesenchymal stem cells as an intravenous infusion once in Phase I clinical trial.

SUMMARY:
This study aims to evaluate safety in subjects with over moderately subacute and chronic atopic dermatitis after an intravenous injection of ADSTEM Inj. Since this is an observational study of patients participated in Phase 1 clinical trials, no drug is administered in this study.

DETAILED DESCRIPTION:
Participants will be followed-up for adverse events on each visit. Visits will be on 6, 12, 18, 24, 30, 36, 48, 60months after treatment of ADSTEM Inj.

Time perspective is both retrospective and prospective.

ELIGIBILITY:
Inclusion Criteria:

* Patients who participated in Phase I clinical trials
* Patients who voluntarily agreed to participate in the study

Exclusion Criteria:

* Patients who can not follow-up from the end of the phase 1 clinical trial to the end of the study

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who participated in Phase I clinical trials
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2022-08-17 (Actual); Study Completion 2022-09-27 (Actual)

PRIMARY OUTCOMES:
Tumor formation | 60months after treatment of ADSTEM Inj.
  The number of subjects with treatment-related tumor formation

SECONDARY OUTCOMES:
Adverse events | 60months after treatment of ADSTEM Inj.
  The number of subjects with treatment-related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Young-joon Seo, M.D, Ph.D, Principal Investigator — Chungnam National University Hospital
Locations (1):
- Chungnam National University Hospital, Daejeon, Chungcheongnam-do, South Korea

IPD SHARING:
Plan to Share IPD: No